CLINICAL TRIAL: NCT03928847
Title: Fibroblast Specific Inhibition of LOXL2 and TGFbeta1 Signaling in Patients With Pulmonary Fibrosis.
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Hal Chapman (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor-Investigator, Hal Chapman, professor, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 17-23008; R01HL142265 (NIH)
Record Dates: First submitted 2019-04-18; First posted 2019-04-26 (Actual); Results first posted 2022-12-22 (Actual); Last update posted 2022-12-22 (Actual); Status verified 2022-12

CONDITIONS: Idiopathic Pulmonary Fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis | interventions — epigallocatechin gallate

STUDY DESIGN:
Masking Description: Open Label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- EGCG PK in healthy volunteers 450 mg (Other): Healthy volunteers: 450 mg Epigallocatechin-3-gallate (EGCG) capsules administered once daily by mouth
  Interventions: Drug: Epigallocatechin-3-gallate (EGCG)
- EGCG PK in healthy volunteers 600 mg (Other): Healthy volunteers: 600 mg Epigallocatechin-3-gallate (EGCG) capsules administered once daily by mouth
  Interventions: Drug: Epigallocatechin-3-gallate (EGCG)
- EGCG PK in healthy volunteers 750 mg (Other): Healthy volunteers: 750 mg Epigallocatechin-3-gallate (EGCG) capsules administered once daily by mouth
  Interventions: Drug: Epigallocatechin-3-gallate (EGCG)
- No treatment control in ILD patients (No Intervention): Patients: not treated with EGCG
- EGCG treatment in ILD patients (Experimental): Patients: 600 mg EGCG capsules once daily by mouth for two weeks
  Interventions: Drug: Epigallocatechin-3-gallate (EGCG)

INTERVENTIONS:
Drug: Epigallocatechin-3-gallate (EGCG) — Epigallocatechin-3-gallate (EGCG) capsules
  Other Names: Teavigo
  Arms: EGCG PK in healthy volunteers 450 mg; EGCG PK in healthy volunteers 600 mg; EGCG PK in healthy volunteers 750 mg; EGCG treatment in ILD patients

SUMMARY:
This is a two part study. In the first part, the pharmacokinetic profile of Epigallocatechin-3-gallate (EGCG) in normal human volunteers given a single oral dose will be determined to set the dose for the second part of the study. In the second part of this study, lung biopsy fragments and urine samples from patients with interstitial lung disease treated with EGCG will be evaluated in biochemical assays and compared to samples from untreated control patients.

DETAILED DESCRIPTION:
This is an interventional study intended to test inhibition of a signaling pathway in vivo in patients with interstitial lung disease, but not intended to affect lung function or disease modifications. Doses of oral Epigallocatechin-3-gallate (EGCG) that achieve plasma levels known to be safe in human volunteers and likely to target fibroblast TGFbeta RI kinase will be established. Disposable fragments of biopsies will be evaluated in biochemical assays including pSmad3 and Snail 1 or assayed to determine lysyl oxidase-like 2 (LOXL2) protein and LOXL2 enzyme activity. Urine collected before and after EGCG exposure will be used to determine whether terminal collagen cross-link breakdown products, termed pyridinoline/deoxypyridinoline (PYD/DPD) are changed from baseline. Blood collected before and after EGCG exposure will be assayed for serum biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Part 1: healthy volunteers
* Part 2:
* study will consist of patients presenting to the UCSF interstitial lung disease (ILD) outpatient clinic with imaging indicative of lung fibrosis but of uncertain classification, and who are willing to take EGCG for a minimum of 2 weeks prior to surgery.

Exclusion Criteria:

* co-morbidities affect hepatic function, such as HCV infection, cirrhosis, or
* using drugs with significant hepatic toxicities

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hal A Chapman, MD, Principal Investigator — UC San Francisco
Locations (1):
- UC San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wei Y, Dong W, Jackson J, Ho TC, Le Saux CJ, Brumwell A, Li X, Klesney-Tait J, Cohen ML, Wolters PJ, Chapman HA. Blocking LOXL2 and TGFbeta1 signalling induces collagen I turnover in precision-cut lung slices derived from patients with idiopathic pulmonary fibrosis. Thorax. 2021 Jul;76(7):729-732. doi: 10.1136/thoraxjnl-2020-215745. Epub 2021 Jan 20. PMID 33472968
- [Result] Chapman HA, Wei Y, Montas G, Leong D, Golden JA, Trinh BN, Wolters PJ, Le Saux CJ, Jones KD, Hills NK, Foster E, Oldham JM, Linderholm AL, Kotak P, Decaris M, Turner S, Song JW. Reversal of TGFbeta1-Driven Profibrotic State in Patients with Pulmonary Fibrosis. N Engl J Med. 2020 Mar 12;382(11):1068-1070. doi: 10.1056/NEJMc1915189. No abstract available. PMID 32160670

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Healthy volunteer recruitment started in 12/1/2017 and ended in 3/30/2018. Subjects were recruited from UCSF community. Advertisements were posted around the campus.
  Patients recruitment started in 6/1/2018 and ended in 12/20/2018. Subjects were recruited from UCSF and UC Davis ILD clinics.
Groups:
- EGCG PK in Healthy Volunteers 450 mg: Teavigo EGCG capsule containing 94% EGCG, 150 mg EGCG/capsule
  Healthy volunteers: 450 mg Epigallocatechin-3-gallate (EGCG) capsules administered once daily by mouth (3 capsules)
- EGCG PK in Healthy Volunteers 600 mg: Teavigo EGCG capsule containing 94% EGCG, 150 mg EGCG/capsule
  Healthy volunteers: 600 mg Epigallocatechin-3-gallate (EGCG) capsules administered once daily by mouth (3 capsules)
- EGCG PK in Healthy Volunteers 750 mg: Teavigo EGCG capsule containing 94% EGCG, 150 mg EGCG/capsule
  Healthy volunteers: 750 mg Epigallocatechin-3-gallate (EGCG) capsules administered once daily by mouth (3 capsules)
- No Treatment Control in ILD Patients: None EGCG treated control ILD patients
- EGCG Treatment in ILD Patients: Teavigo EGCG capsule containing 94% EGCG, 150 mg EGCG/capsule
  Patients: 600 mg EGCG capsules once daily by mouth for two weeks (4 capsules once daily)
Period: Overall Study
Arm/Group | EGCG PK in Healthy Volunteers 450 mg | EGCG PK in Healthy Volunteers 600 mg | EGCG PK in Healthy Volunteers 750 mg | No Treatment Control in ILD Patients | EGCG Treatment in ILD Patients
Started | 5 | 5 | 5 | 10 | 10
Completed | 5 | 5 | 5 | 10 | 10
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- EGCG PK in Healthy Volunteers 450 mg: Healthy volunteers: 450 mg Epigallocatechin-3-gallate (EGCG) capsules administered once daily by mouth
  Epigallocatechin-3-gallate (EGCG): 3 EGCG capsules
- EGCG PK in Healthy Volunteers 600 mg: Healthy volunteers: 600 mg Epigallocatechin-3-gallate (EGCG) capsules administered once daily by mouth
  Epigallocatechin-3-gallate (EGCG): 4 EGCG capsules
- EGCG PK in Healthy Volunteers 750 mg: Healthy volunteers: 750 mg Epigallocatechin-3-gallate (EGCG) capsules administered once daily by mouth
  Epigallocatechin-3-gallate (EGCG): 5 EGCG capsules
- No Treatment Control in ILD Patients: ILD patients that were not treated with EGCG are used as controls.
- EGCG Treatment in ILD Patients: Patients: 600 mg EGCG capsules once daily by mouth for two weeks
  Epigallocatechin-3-gallate (EGCG): 4 EGCG capsules
- Total: Total of all reporting groups
Arm/Group | EGCG PK in Healthy Volunteers 450 mg | EGCG PK in Healthy Volunteers 600 mg | EGCG PK in Healthy Volunteers 750 mg | No Treatment Control in ILD Patients | EGCG Treatment in ILD Patients | Total
Number analyzed (Participants) | 5 | 5 | 5 | 10 | 10 | 35
Age, Customized [Median (Full Range); unit: years] | 64 [55 to 69] | 62 [45 to 67] | 68 [53 to 70] | 64 [56 to 71] | 65 [58 to 70] | 64 [45 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 3 | 5 | 6 | 20
  Male | 2 | 2 | 2 | 5 | 4 | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 3 | 2 | 2 | 4 | 1 | 12
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0
  White | 2 | 3 | 3 | 6 | 9 | 23
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 | 5 | 5 | 6 | 10 | 31
  South Korea | 0 | 0 | 0 | 4 | 0 | 4
High-resolution computed tomography (HRCT) imaging indicative of lung fibrosis [Count of Participants; unit: Participants] | 0 | 0 | 0 | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: EGCG PK Level in Healthy Volunteers
Description: EGCG plasma levels in healthy volunteers were measured at 0, 0.5, 2, and 4 hours after a single dose at 450 mg, 600 mg, or 750 mg dosage by liquid chromatography-mass spectrometry (LC-MS).
Time Frame: 0, 0.5, 2, 4 hours after EGCG
Measure: Mean (Standard Deviation); unit: nM
Groups:
- EGCG PK in Healthy Volunteers 450 mg: Teavigo EGCG capsule containing 94% EGCG, 150 mg EGCG/capsule
  Healthy volunteers: 450 mg Epigallocatechin-3-gallate (EGCG) capsules administered once daily by mouth
- ECGC PK in Healthy Volunteers 600 mg: Teavigo EGCG capsule containing 94% EGCG, 150 mg EGCG/capsule
  Healthy volunteers: 600 mg Epigallocatechin-3-gallate (EGCG) capsules administered once daily by mouth
- EGCG PK in Healthy Volunteers 750 mg: Teavigo EGCG capsule containing 94% EGCG, 150 mg EGCG/capsule
  Healthy volunteers: 750 mg Epigallocatechin-3-gallate (EGCG) capsules administered once daily by mouth
Arm/Group | EGCG PK in Healthy Volunteers 450 mg | ECGC PK in Healthy Volunteers 600 mg | EGCG PK in Healthy Volunteers 750 mg
Number analyzed (Participants) | 5 | 5 | 5
nM
  0 hour after EGCG | NA (NA) — below the level of detection | NA (NA) — below the level of detection | NA (NA) — below the level of detection
  0.5 hour after EGCG | 861 (761) | 612 (531) | 3126 (4159)
  2 hours after EGCG | 1136 (666) | 2266 (2174) | 1582 (536)
  4 hours after EGCG | 659 (640) | 741 (226) | 702 (293)
Statistical Analysis 1: Comparison: EGCG PK in Healthy Volunteers 450 mg vs ECGC PK in Healthy Volunteers 600 mg vs EGCG PK in Healthy Volunteers 750 mg; Test type: Superiority — The mean EGCG blood levels were compared among 450 mg, 600 mg, and 750 mg groups; Mean Difference (Net) = 250

2. Primary Outcome: Change of Serum Biomarker COMP Before and After EGCG Treatment in ILD Patients
Description: Change from baseline to day 14 in serum biomarkers associated with IPF, Cartilage Oligomeric Matrix Protein (COMP) measured by ELISA.
Time Frame: Day 1 to day 14
Population: Serum biomarker COMP was measured by ELISA and compared before and after EGCG treatment.
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | EGCG Treatment in ILD Patients
Number analyzed (Participants) | 10
ng/ml
  Before EGCG treatment | 137.2 (53.8)
  After EGCG treatment | 97.9 (26.9)
Statistical Analysis 1: Comparison: EGCG Treatment in ILD Patients; Test type: Other — ELISA data from each patient before and after EGCG treatment were compared and analyzed with the use of the Wilcoxon signed-rank test (two-tailed); p < 0.01, Wilcoxon (Mann-Whitney)

3. Primary Outcome: Change of Serum Biomarker Periostin Before and After EGCG Treatment in ILD Patients
Description: Change from baseline to day 14 in serum biomarkers associated with IPF, Periostin measured by ELISA.
Time Frame: Day 1 to day 14
Population: Serum biomarker Periostin was measured by ELISA and compared before and after EGCG treatment.
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | EGCG Treatment in ILD Patients
Number analyzed (Participants) | 10
ng/ml
  Before EGCG treatment | 41.9 (15.9)
  After EGCG treatment | 35.2 (11.7)
Statistical Analysis 1: Comparison: EGCG Treatment in ILD Patients; Test type: Other — [test comment as in outcome 2, analysis 1]; p < 0.01, Wilcoxon (Mann-Whitney)

4. Primary Outcome: Difference of Biomarker Snail1 Between EGCG-treated and Non-treated Patient Groups
Description: Levels of biomarker Snail1 in lung biopsy tissues 14 days after EGCG were measured by western blot and differences were compared between EGCG-treated and non-treated groups.
Time Frame: 14 days
Measure: Mean (Standard Deviation); unit: percentage of reference sample
Arm/Group | No Treatment Control in ILD Patients | EGCG Treatment in ILD Patients
Number analyzed (Participants) | 10 | 10
percentage of reference sample | 0.825 (0.332) | 0.132 (0.098)
Statistical Analysis 1: Comparison: No Treatment Control in ILD Patients vs EGCG Treatment in ILD Patients; Test type: Other; p < 0.01, Kruskal-Wallis

5. Primary Outcome: Difference of Biomarker Collagen I Between EGCG-treated and Non-treated Patient Groups
Description: Levels of biomarker Collagen I in lung biopsy tissues 14 days after EGCG were measured by western blot and differences were compared between EGCG-treated and non-treated groups.
Time Frame: 14 days
Measure: Mean (Standard Deviation); unit: percentage of reference sample
Arm/Group | No Treatment Control in ILD Patients | EGCG Treatment in ILD Patients
Number analyzed (Participants) | 10 | 10
percentage of reference sample | 0.894 (0.375) | 0.136 (0.058)
Statistical Analysis 1: Comparison: EGCG Treatment in ILD Patients; Test type: Other; p < 0.01, Kruskal-Wallis

6. Primary Outcome: Difference of Biomarker p-Smad3 Between EGCG-treated and Non-treated Patient Groups
Description: Levels of biomarker p-Smad3 in lung biopsy tissues 14 days after EGCG were measured by western blot and differences were compared between EGCG-treated and non-treated groups.
Time Frame: 14 days
Measure: Mean (Standard Deviation); unit: percentage of reference sample
Arm/Group | No Treatment Control in ILD Patients | EGCG Treatment in ILD Patients
Number analyzed (Participants) | 10 | 10
percentage of reference sample | 0.913 (0.201) | 0.284 (0.126)
Statistical Analysis 1: Comparison: No Treatment Control in ILD Patients vs EGCG Treatment in ILD Patients; Test type: Other; p < 0.01, Kruskal-Wallis

ADVERSE EVENTS:
Time Frame: Adverse event data were collected during the whole course of the study (14 days).
Groups:
- EGCG PK in Healthy Volunteers 600 mg: Teavigo EGCG capsule containing 94% EGCG, 150 mg EGCG/capsule
  Healthy volunteers: 600 mg Epigallocatechin-3-gallate (EGCG) capsules administered once daily by mouth
Arm/Group | EGCG PK in Healthy Volunteers 450 mg | EGCG PK in Healthy Volunteers 600 mg | EGCG PK in Healthy Volunteers 750 mg | No Treatment Control in ILD Patients | EGCG Treatment in ILD Patients
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5 | 0/5 | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5 | 0/5 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/5 | 0/5 | 0/5 | 0/10 | 0/10

LIMITATIONS AND CAVEATS:
The study was a pilot study with a small sample size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2018-01-30): https://cdn.clinicaltrials.gov/large-docs/47/NCT03928847/Prot_SAP_000.pdf
  • Informed Consent Form: Consent Form for ILD Patients (2018-01-30): https://cdn.clinicaltrials.gov/large-docs/47/NCT03928847/ICF_001.pdf
  • Informed Consent Form: Consent Form for Healthy Volunteers (2018-01-30): https://cdn.clinicaltrials.gov/large-docs/47/NCT03928847/ICF_002.pdf